CLINICAL TRIAL: NCT03661281
Title: Function Following Thumb MP Fusion and IP Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-01281
Record Dates: First submitted 2018-08-09; First posted 2018-09-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Pinch Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulated Thumb Arthrodesis (Experimental): Subjects will have their thumb immobilized in 2 prefabricated wrist splints to simulate 2 different fusion positions tested: one splint to simulate the MCP fusion and one to represent the IP fusion. Patients will complete hand function tests in each of the splints to evaluate hand function.
  Interventions: Diagnostic Test: Jebsen Taylor Hand function test; Diagnostic Test: Pinch strength; Diagnostic Test: Grooved pegboard test

INTERVENTIONS:
Diagnostic Test: Jebsen Taylor Hand function test — consists of seven test items, which are felt to represent various hand activities. These test items include: writing a short sentence; turning over 365 inch cards; picking up small objects and placing in a container; stacking checkers; simulated eating; moving empty large cans; and moving weighted large cans.
Diagnostic Test: Pinch strength — Measured in every splint position using a standard dynamometer
Diagnostic Test: Grooved pegboard test — Time will be measured and compared between control, MP splint and IP splint

SUMMARY:
This study is to determine function following simulated thumb metacarpophalangeal (MP) and thumb interphalangeal (IP) joint fusion. The investigators want to determine the functional limitation created by MP and IP joint fusion. 20-30 volunteers will be fitted for custom molded orthoplast splints immobilizing either the MP or IP joint. The volunteers will then be taken through multiple tests including lateral pinch strength, tip pinch, grip strength, grooved pegboard test time, and Jebson Taylor test. Each patient will be tested without a splint, with their MP joint immobilized and with their IP joint immobilized. The results of this study can be used for patient education before surgery in order to help them make informed decisions as well as manage expectations. It can also serve as a decision aid in pinch restoration in the context of ulnar nerve palsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a healthy volunteer
* Patient is willing and able to review and sign a study informed consent form

Exclusion Criteria:

* Any subject who does not want to voluntarily participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Jebsen Taylor hand function test | 1 Month
  This consists of seven test items, which are felt to represent various hand activities. Each activity will be timed.

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Melamed, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided